CLINICAL TRIAL: NCT03388775
Title: Real World Study of Deep Venous Thrombosis in Brazil. Analysis of Prospective Cases in University Hospitals in the State of São Paulo
Brief Title: Real World Study of Deep Venous Thrombosis. Analysis of Prospective Cases in University Hospitals of São Paulo
Acronym: DVT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundação Faculdade Regional de Medicina de São José do Rio Preto (Other)
Collaborators: University of Ribeirao Preto (Other)
Responsible Party: Principal Investigator, Selma Regina de Oliveira Raymundo, Principal Investigator, Fundação Faculdade Regional de Medicina de São José do Rio Preto
Other Study IDs: DVT 2017
Record Dates: First submitted 2017-10-31; First posted 2018-01-03 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2023-12

CONDITIONS: Registry
Keywords: deep vein thrombosis; assessment; risk factors
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with deep venous thrombosis: Five-year prospective records of deep venous thrombosis have been collected by the RHEUNI group of five public schools in the State of São Paulo.
  Demographic data of patients will be evaluated along with the main risk factors, clinical picture, diagnostic methods, use of different drugs to treat the disease and its complications.
  Interventions: Other: deep venous thrombosis

INTERVENTIONS:
Other: deep venous thrombosis — Five-year prospective analysis of deep venous thrombosis performed by the RHEUNI group of five public schools in the State of São Paulo.

SUMMARY:
Background: Deep venous thrombosis (DVT) is a common and important vascular disease due to its morbidity and mortality.

Its incidence remains high throughout the world and constitutes serious problems for national and international public health.

Several inherited and/or acquired risk factors may be responsible for thrombus formation. Few epidemiological data regarding real world panorama of this disease in South America and Brazil is available in the literature.

Objective: Evaluate demographic data, diagnostic methods and treatment of deep vein thrombosis in the real world in public university hospitals in Brazil.

Methods: Five-year prospective records of deep venous thrombosis have been collected by the RHEUNI group of five public schools in the State of São Paulo.

Demographic data of patients will be evaluated along with the main risk factors, clinical picture, diagnostic methods, use of different drugs to treat the disease and its complications. Digital platform has been used in data collection. Is a multicenter study and analysis will be performed using Microsoft Excel and Epi-Info.

Key words: deep vein thrombosis, assessment, risk factors, demographic data.

DETAILED DESCRIPTION:
Introduction DVT is a multidisciplinary disease, mainly as consequence of surgical or clinical conditions, and the acute pulmonary embolism and the post-thrombotic syndrome (PTS) are the most serious complications.

The incidence of deep venous thrombosis of the lower limbs in the population is from 0.2 to 0.7 cases per 1,000 inhabitants/year and in Brazil an estimated incidence of 0.6 cases/1000 inhabitants/year has been estimated.

Risk factors for DVT include: advanced age, history of immobilization or prolonged bed rest during hospitalization, obesity, smoking, recent surgery, previous VTE episodes, cancer, major or lower limb trauma, cancer therapy, acute infectious disease, heart failure, respiratory insufficiency, contraceptive use or hormone replacement therapy, pregnancy or postpartum, stroke with motor deficit, family history of VTE (thrombophilia).

The clinical diagnosis of DVT, based on physical examination only, is imprecise and insensitive and only one-third or less of the clinical suspicions are confirmed by imaging tests.

The primary goals of DVT treatment are to prevent and / or treat their complications. Anticoagulant therapy is efficacious but associated to some risk of bleeding. Mechanical prophylactic measures (ambulation and use of elastic stockings with gradual compression) are important in high risk patients and in cases with contraindication of anticoagulants.

Although well known, epidemiological data on this disease may have some particularities related to geographic regions. Data from registries in USA and Europe has shown some differences in demographic profile, risk factors and treatments.

Few epidemiological data regarding real world panorama of this disease in South America and Brazil is available in the literature.

So, the objective of this was to evaluate demographic data, diagnostic methods and and treatment of deep vein thrombosis in the real world in public university hospitals in Brazil.

Methods

1. Population of patients The Registries of the Universities Hospitals (RHEUNI) in Brazil have been registry consecutive patients with deep venous thrombosis that was started on July 2013, with a prospective collection of epidemiological data of patients referred to five public university hospitals in the state of São Paulo (Base Hospital of São José do Rio Preto Medical School , Clinics Hospital Ribeirão Preto Medical School of São Paulo University, Clinics Hospital of Campinas University, Clinics Hospital of Botucatu Medical School of the Paulista State University, Clinics Hospital of Marília Medical School). This study was approved in the ethics committees of all institutions. An informed consent form was signed by the patient after explaining the purpose of the study.

   Inclusion criteria are as follows: patients with venous thrombosis in any site, male or female, regardless of age, with first episode or recurrent episodes and with or without pulmonary embolism.

   There are no exclusion criteria.
2. Patients registration Patients has been performed in planned digital spreadsheets and loaded in a computer program for statistical analysis (Epi-Info). Every single completed worksheets will be exported to Excel worksheet for statistical analysis.

   The main outcomes to be reviewed are: demographic characteristics (age, sex and color), main risk factors for DVT and time of clinical history collected from consecutive patients referred for those Hospitals. The main symptoms and signs reported by patients, the sectors affected by thrombosis, as well as the diagnostic tools employed were registered.
3. Worksheet form The recorded characteristics and backgrounds of patients with venous thrombosis include: age, gender, and main clinics or surgical risk factors. In addition, the main signs and symptoms and the sectors affected by thrombosis will be reported, and the diagnostic tools employed.

   The use of various anticoagulants for the treatment of venous thrombosis and complications related mainly to bleeding will be analyzed.
4. Responsibilities of researchers and institutions The principal investigators and co-participants are committed to maintain the project along time with accurate information and to participate in quarterly meetings of the RHEUNI group to analyze the progress of the project and to publish the results.

   The project has no external financial support and there is no conflicts of interest of any researcher.
5. Statistical analysis The analyzes will include the sociodemographic characteristics of patients with deep venous thrombosis. The projected number of cases during the study period is approximately 800 patients. All analyzes will be conducted using Microsoft Excel.

The objective of the study is to evaluate the demographic data and the most common clinical characteristics of patients with deep venous thrombosis in public hospitals, their main predisposing factors, the most commonly used diagnostic tests and the treatments performed. The participating hospitals have common characteristics: they are large public university hospitals with a significant number of patients hospitalized and trained by new angiologists and vascular surgeons in the Sao Paulo State. This study will represent a significant sample of deep venous thrombosis and its main risk factors and treatments performed so that this disease can be prevented in some hospital and post-discharge situations in an attempt to reduce its incidence. Treatment in our real world in most cases is not possible to be performed outpatient initially due to socio-economic conditions of patients and difficulty in acquiring the new oral anticoagulants.

ELIGIBILITY:
Inclusion Criteria:

* patients with venous thrombosis in any site, male or female, regardless of age, with first episode or recurrent episodes and with or without pulmonary embolism.

Exclusion Criteria:

* There are no exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with venous thrombosis in any site, male or female, regardless of age, with first episode or recurrent episodes and with or without pulmonar embolism.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2013-07 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of risk factors for DVT | Five Years
  1. Inheriting a blood-clotting disorder.
  2. Prolonged bed rest, such as during a long hospital stay, or paralysis.
  3. Injury or surgery.
  4. Pregnancy.
  5. Birth control pills (oral contraceptives) or hormone replacement therapy.
  6. Being overweight or obese.
  7. Smoking.
  8. Cancer.
  9. Heart failure.
  10. Inflammatory bowel disease.
  11. A personal or family history of deep vein thrombosis or pulmonary embolism.
  12. Age. Being older than 60 increases your risk of DVT.

SECONDARY OUTCOMES:
Types of treatment performed in the real world | Five Years
  Anticoagulation.
  Types of treatment performed in the real world
  Description:
  Anticoagulation.
  * Unfractionated heparin, which is given into a vein (intravenously) - This may be the preferred choice in certain circumstances, such as if the patient has severe kidney failure or unstable blood pressure.
  * Direct oral anticoagulants - These are available in pill form; they include rivaroxaban (brand name: Xarelto) and apixaban (brand name: Eliquis).
  The choice of anticoagulant depends upon multiple factors, including the preference of the patient and the healthcare provider, the patient's medical history and other conditions, and cost considerations.

CONTACTS AND LOCATIONS:
Overall Officials: Selma R Raymundo, MD; PhD, Principal Investigator — Fundação Faculdade Regional de Medicina de São Jose Do Rio Preto
Locations (1):
- Clinics Hospital of Faculty of Medicine of Paulista State University, Botucatu, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No